CLINICAL TRIAL: NCT01407926
Title: The Effects of a Nurse-Led Interprofessional Mental Health Promotion Intervention Among Older Home Care Clients
Brief Title: Nurse-Led Interprofessional Mental Health Promotion Intervention for Older Home Care Clients
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHE-101531; 06510 (Other Grant/Funding Number: Ontario Ministry of Health and Long-Term Care)
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Depressive Symptoms
Keywords: Depression; Aging; Clinical Effectiveness; Home Care; Nurse-Led
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nurse-Led Mental Health Promotion Group: Interprofessional nurse-led strategy involving regular home visits over 6 months by an RN and PSW. The RN will conduct a comprehensive health assessment and screen clients for risk factors for depression and other chronic conditions, implement health promotion strategies to address this risk factors and enhance health, review their medications, conduct in-home exercise , refer clients to other health services
  Interventions: Other: Nurse-Led Mental Health Promotion Intervention

INTERVENTIONS:
Other: Nurse-Led Mental Health Promotion Intervention — The nurse-led intervention is a multi-faceted 6-month program led by a Registered Nurse that involves regular home visits, monthly case conferences, and evidence-based assessment and management of depression using an interprofessional approach.

SUMMARY:
Objective: The objective of this study is to evaluate the feasibility, acceptability and effectiveness of a 6-month nurse-led, interprofessional mental health promotion intervention aimed at older home care clients with depressive symptoms using personal support services.

Methods/Design: This one-group pre-test post-test study aims to recruit a total of 250 long-stay (> 60 days) home care clients, 70 years or older, with depressive symptoms who are receiving personal support services through a home care program in Ontario, Canada. The nurse-led intervention is a multi-faceted 6-month program led by a Registered Nurse that involves regular home visits, monthly case conferences, and evidence-based assessment and management of depression using an interprofessional approach. The primary outcome is the change in severity of depressive symptoms from baseline to 6 months using the Centre for Epidemiological Studies in Depression Scale. Secondary outcomes include changes in the prevalence of depressive symptoms and anxiety, health-related quality of life, cognitive function, and the rate and appropriateness of depression treatment from baseline to 12 months. Changes in the costs of use of health services will be assessed from a societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* long-stay (> 60 days) home care clients
* 70 years or older
* newly referred to and receiving PSS through the CCAC
* living in the community (not in a long-term care home)
* mentally competent to give informed consent (or with a substitute decision-maker available)
* competent in English (or with an interpreter available)
* screens positive for depressive symptoms

Exclusion Criteria:

* receiving palliative care services
* not competent in English and no interpreter available
* not mentally competent to give informed consent and no substitute decision-maker available

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older home care clients receiving personal support services through a home care program in Southern Ontario
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen F Markle-Reid, RN, PhD, Principal Investigator — McMaster University, School of Nursing
Locations (1):
- McMaster University, School of Nursing, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Markle-Reid M, McAiney C, Forbes D, Thabane L, Gibson M, Browne G, Hoch JS, Peirce T, Busing B. An interprofessional nurse-led mental health promotion intervention for older home care clients with depressive symptoms. BMC Geriatr. 2014 May 10;14:62. doi: 10.1186/1471-2318-14-62. PMID 24886344
- [Derived] Markle-Reid MF, McAiney C, Forbes D, Thabane L, Gibson M, Hoch JS, Browne G, Peirce T, Busing B. Reducing depression in older home care clients: design of a prospective study of a nurse-led interprofessional mental health promotion intervention. BMC Geriatr. 2011 Aug 25;11:50. doi: 10.1186/1471-2318-11-50. PMID 21867539

RESULTS

PARTICIPANT FLOW:
Groups:
- Nurse-Led Mental Health Promotion Group: Interprofessional nurse-led strategy involving regular home visits over 6 months by an RN and PSW. The RN will conduct a comprehensive health assessment and screen clients for risk factors for depression and other chronic conditions, implement health promotion strategies to address this risk factors and enhance health, review their medications, conduct in-home exercise , refer clients to other health services
  Nurse-Led Mental Health Promotion Intervention : The nurse-led intervention is a multi-faceted 6-month program led by a Registered Nurse that involves regular home visits, monthly case conferences, and evidence-based assessment and management of depression using an interprofessional approach.
Period: Overall Study
Arm/Group | Nurse-Led Mental Health Promotion Group
Started | 142
Completed | 87
Not Completed | 55
Not completed — Lost to Follow-up | 55

BASELINE CHARACTERISTICS:
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 82 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 50
Region of Enrollment [Number; unit: participants]
  Canada | 142

OUTCOME MEASURES:

1. Primary Outcome: Centre for Epidemiological Studies in Depression Scale
Description: The CES-D consists of 20 items, which range from 0-60, with higher scores indicating greater severity of depressive symptoms. It has been used in prior randomized controlled trials by three of the study investigators that involved older home care clients with mood disorders and has a high degree of reliability, content, construct and criterion related validity, distinguishes between depressed and non-depressed people, and is a sensitive tool for measuring changes in depressive symptoms over time in psychiatric populations.
Time Frame: Baseline to 12 months
Population: 12 months minus baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 79
units on a scale | -3.52 [-5.77 to -1.27]

2. Secondary Outcome: Generalized Anxiety Disorder Screener
Description: The Generalised Anxiety Disorder Assessment (GAD-7) is a seven item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day".
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions.
  GAD-7 total score for the seven items ranges from 0 to 21. Scores represent:
  * 0-5 = Mild anxiety
  * 6-10 = Moderate anxiety
  * 11-15 = Moderately severe anxiety
  * 15-21 = Severe anxiety
  When used as a screening tool, further evaluation is recommended when the score is 10 or greater
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | -1.83 [-3.03 to -0.62]

3. Secondary Outcome: SF-12 Physical Composite Index
Description: The SF-12 is a multipurpose short form to measure health status. There are 10 domains: Physical Composite Index (score range from 0-100); Physical Functioning Index (score range from 0-100); Role Limitation Physical Index (score range 0-100); Pain Index Score (score range from 0-100); General Health Index (score range from 0-100); Mental Health Composite Index (score range from 1-100); Vitality Index (score range from 0-100); Social Functioning Index (score rang 0-100); Role Limitation Emotional Index (score range 0-100); and SF-12 Mental Health Index (score range from 0-100), the higher the score means a better outcome
Time Frame: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 8.70 [3.65 to 13.75]

4. Secondary Outcome: SF-12 Physical Functioning Index
Description: The SF-12 is a multipurpose short form to measure health status. There are 10 domains: Physical Composite Index (score range from 0-100); Physical Functioning Index (score range from 0-100); Role Limitation Physical Index (score range 0-100); Pain Index Score (score range from 0-100); General Health Index (score range from 0-100); Mental Health Composite Index (score range from 1-100); Vitality Index (score range from 0-100); Social Functioning Index (score rang 0-100); Role Limitation Emotional Index (score range 0-100); and SF-12 Mental Health Index (score range from 0-100), the higher the score means the better the outcome.
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 6.88 [-0.37 to 14.12]

5. Secondary Outcome: SF-12 Role Limitation Physical Index
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 15.47 [6.87 to 24.07]

6. Secondary Outcome: SF-12 Pain Index Score
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 5.94 [-3.10 to 14.98]

7. Secondary Outcome: SF-12 General Health Index
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | -0.25 [-6.31 to 5.81]

8. Secondary Outcome: SF-12 Mental Health Composite Index
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 8.96 [3.69 to 14.23]

9. Secondary Outcome: SF-12 Vitality Index Score
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 8.75 [0.39 to 17.11]

10. Secondary Outcome: SF-12 Social Functioning Index
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 4.38 [-8.57 to 17.32]

11. Secondary Outcome: SF-12 Role Limitation Emotional Index
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 10.31 [1.09 to 19.53]

12. Secondary Outcome: SF-12 Mental Health Index
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: 12 months minus Baseline value
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse-Led Mental Health Promotion Group
Number analyzed (Participants) | 80
units on a scale | 10.00 [3.53 to 16.47]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Nurse-Led Mental Health Promotion Group
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes